CLINICAL TRIAL: NCT02980484
Title: fMRI-neuronavigated Repetitive Transcranial Magnetic Stimulation for the Treatment of Major Depression Associated With Traumatic Brain Injury
Brief Title: fMRI-neuronavigated rTMS for the Treatment of Major Depression Associated With TBI
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigators left the institution for unrelated reasons
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201603051
Record Dates: First submitted 2016-02-25; First posted 2016-12-02 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Major Depressive Disorder; Traumatic Brain Injury
Keywords: rTMS
MeSH Terms: conditions — Depressive Disorder, Major; Brain Injuries, Traumatic | interventions — Exercise; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Randomized double-blind sham-controlled trial with an optional open-label crossover extension for subjects randomized to sham group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active rTMS (Experimental): Subjects will receive a full course of 20 rTMS treatments over 20 consecutive weekdays as described above.
  Interventions: Procedure: Active
- Sham/crossover rTMS (Sham Comparator): Rather than receiving active treatment, subjects will receive sham treatment designed to be indistinguishable from active treatment to the patient. After completion of the sham course, patients will have the option to receive open-label active treatment at no cost.
  Interventions: Procedure: Sham

INTERVENTIONS:
Procedure: Active — Repetitive transcranial magnetic stimulation (rTMS) will be applied to the left dorsolateral prefrontal cortex (DLPFC) (4000 pulses, 10 Hz, 5-sec trains, 25-sec inter-train interval) followed by the right DLPFC (1000 pulses, 1 Hz frequency, single train). The DLPFC will be identified using individual subject-level resting-state network estimation (Hacker et al, 2013). Each treatment will be completed over the course of 1 hour, and each subject will receive a total of 20 treatments over the course of 20 consecutive weekdays.
  Arms: Active rTMS
Procedure: Sham — Treatment that looks and feels similar to active rTMS will be administered as a sham treatment.
  Arms: Sham/crossover rTMS

SUMMARY:
This pilot study aims to investigate the efficacy of fMRI-targeted repetitive transcranial magnetic stimulation (rTMS) in treatment of major depression associated with traumatic brain injury (TBI). Half of patients will receive active treatment, while the other will receive a sham treatment with the option of receiving open-label active treatment afterwards.

DETAILED DESCRIPTION:
rTMS is an FDA-approved treatment for major depressive disorder, but its utility has not yet been investigated for major depression associated with traumatic brain injury.

This will be a prospective double-blind randomized sham-controlled crossover study. Patients in the treatment group will receive 20 sessions of high-frequency rTMS over the left dorsolateral prefrontal cortex (DLPFC) and low-frequency rTMS over the right DLPFC. The DLPFC will be identified as target by using individual subject-level resting state network estimation (Hacker et al, 2013). Patients in the control group will receive 20 sham treatments designed to be visibly indistinguishable from active treatment, and will subsequently have the option to be crossed over to receive active treatment with the aforementioned protocol. A subgroup of patients in each group will receive more detailed diffusion imaging (diffusion tensor and diffusion kurtosis imaging) and resting state fMRI scans before and after the treatment in order to assess for changes in white matter integrity and functional connectivity associated with the treatment.

ELIGIBILITY:
Inclusion criteria:

* Adults age 18 to 65
* History of traumatic brain injury (TBI) at least two weeks prior to study initiation
* Presence of an active major depressive episode as defined by DSM-5 criteria, including depression secondary to traumatic brain injury
* Baseline score of 10 or greater on Montgomery-Asberg Depression Rating Scale (MADRS)
* Failure of at least one prior antidepressant trial after the traumatic brain injury

Exclusion criteria

History of:

* Moderate or severe substance use disorder in the past six months as defined by DSM-5 criteria, with the exception of cannabis and nicotine use disorders.
* Dementia, as defined by treating neurologist
* Moderate or severe autism spectrum disorder
* Bipolar disorder
* Schizophrenia spectrum disorders

Current evidence of:

* Substance-induced mood disorder
* Active psychotic symptoms
* Depression secondary to a general medical illness, with the exception of TBI
* Dysphoria better explained by a baseline personality disorder than a major depressive episode
* Dysphoria better explained by a baseline anxiety disorder (including post-traumatic stress disorder) rather than a major depressive episode
* Active suicidal ideation

Contraindications to rTMS treatment:

* Seizure disorder
* Significantly elevated seizure risk, as determined by clinician assessment
* TBI associated with elevated seizure risk, including penetrating injury and/or cortical intraparenchymal hemorrhage
* Presence of metallic objects within the head
* Presence of an implanted neurostimulation device within the head

Contraindications to MRI

* Severe claustrophobia
* Severe pain/illness exacerbated by lying prone in the scanner
* Presence of non-MRI compatible metal foreign bodies or implants
* Weight in excess of 350 lbs
* Shoulder width in excess of maximum tolerable width for scanner

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Improvement in depressive symptoms | Difference between pre-treatment (baseline) and post-treatment (4 weeks)
  This will be measured as the mean percentage change in baseline scores on Montgomery-Asberg Depression Rating Scale (MADRS) before treatment and immediately after the 4-week treatment period.

SECONDARY OUTCOMES:
Changes in resting-state fMRI and DTI findings | Difference between pre-treatment (baseline) and post-treatment (4 weeks)
  MRI imaging will be conducted to assess resting-state functional connectivity using functional magnetic resonance imaging (fMRI). More detailed structural (DTI) and functional (fMRI) imaging will be measured in a subgroup of patients.
Changes in NIH Toolbox Cognitive, Emotional, and Quality of Life batteries | Difference between pre-treatment (baseline) and post-treatment (4 weeks)
  The NIH Toolbox Cognitive battery will be used to determine change in cognitive symptoms with treatment. Emotional battery and TBI-QoL scales will be used to determine change in general neuropsychiatric symptom burden.
Changes in temperament and character | Difference between pre-treatment (baseline) and post-treatment (4 weeks)
  Will administer the 140-question Temperament and Character Inventory (TCI-R140) before and after treatment.
Response and remission rates in depressive symptoms | Difference between pre-treatment (baseline) and post-treatment (4 weeks)
  Percentage of subjects achieving response (>50% improvement in MADRS) and remission (final MADRS score <7) before treatment and immediately after the 4-week treatment period.
Changes in headache scales | Difference between pre-treatment (baseline) and post-treatment (4 weeks)
  Mean percentage improvement in HIT-6 headache scores
Changes in tinnitus score | Difference between pre-treatment (baseline) and post-treatment (4 weeks)
  Mean percentage improvement in tinnitus severity score and mini-Tinnitus Questionnaire scores

CONTACTS AND LOCATIONS:
Overall Officials: Shan H Siddiqi, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified neuroimaging data will be submitted to FITBIR (Federal Interagency TBI Research)